CLINICAL TRIAL: NCT03513380
Title: Motivational High Intensity Training Through a Cutting-edge Gaming Platform. A Randomised, Controlled Trial
Brief Title: Can Gaming Get You Fit? A High-Intensity Exergaming Intervention in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017/1501
Record Dates: First submitted 2018-04-05; First posted 2018-05-01 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Sedentary Lifestyle
Keywords: Exercise therapy; Physical fitness; Gaming; Adult; Healthy lifestyle; Fitness testing
MeSH Terms: conditions — Sedentary Behavior | interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergaming (Experimental): free access to the exergame PedalTanks
  Interventions: Behavioral: Exergaming
- Control (No Intervention): recommended to continue with their normal daily routine

INTERVENTIONS:
Behavioral: Exergaming — free access to the exergame PedalTanks during 6 months
  Other Names: PlayPulse; PedalTanks
  Arms: Exergaming

SUMMARY:
The purpose of this project is to assess if playing a newly developed videogame that require physical activity (e.g. exergame) can lead to health benefits. The project will include 50 adult participants that are not particularly physically active. They will be randomized into two groups where one group will be given free access to the exergame for 6 months. The physical fitness (maximal oxygen consumption), blood markers of cardiometabolic health and body composition of the subjects will be tested before, mid-ways and after the intervention period. Also, the participants gaming frequency will be registered throughout the 6-month period. Aim of this study is to investigate if access to this game can provide health benefits for individuals who are not motivated to take part in regular physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary (<150 mins of moderate intensity physical activity/week)
* Able to ride a bike for up to 60 minutes

Exclusion Criteria:

* Known cardiovascular disease
* Taking beta-blockers or anti-arrhythmic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
VO2max (Maximal Aerobic Capacity) | 3 months
VO2max (Maximal Aerobic Capacity) | 6 months

SECONDARY OUTCOMES:
Daily average energy expenditure | 3 and 6 months
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period, 3-months and 6-months.
Daily average number of steps | 3 and 6 months
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period, 3-months and 6-months.
Daily time in sedentary activity (< 3.0 metabolic equivalents = METs) | 3 and 6 months
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period, 3-months and 6-months.
Daily time in moderate intensity activity (3.0-6.0 metabolic equivalents = METs) | 3 and 6 months
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period, 3-months and 6-months.
Daily time in vigorous intensity activity (6.0-9.0 metabolic equivalents = METs) | 3 and 6 months
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period, 3-months and 6-months.
Daily time in very vigorous intensity activity (>9.0 metabolic equivalents = METs) | 3 and 6 months
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period, 3-months and 6-months.
Daily average total physical activity duration | 3 and 6 months
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period, 3-months and 6-months.
Bioelectrical impedance | 3 and 6 months
  Body composition assessed using bioelectrical impedance analysis (InBody 720)
Blood Pressure | 3 and 6 months
Fasting circulating glucose, as blood marker of cardiometabolic health | 6 months
Lipid profile, as blood marker of cardiometabolic health | 6 months
Circulating insulin concentration, as blood marker of cardiometabolic health | 6 months
glucose response to a 2 hour glucose tolerance test, as blood marker of cardiometabolic health | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Risa, PhD, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Circulation and Medical Imaging, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Berg J, Wang AI, Lydersen S, Moholdt T. Can Gaming Get You Fit? Front Physiol. 2020 Aug 20;11:1017. doi: 10.3389/fphys.2020.01017. eCollection 2020. PMID 32973553